CLINICAL TRIAL: NCT01504126
Title: Feasibility Study: Therapeutic Targeting of Stress Factors in Ovarian Cancer Patients
Brief Title: Propranolol Hydrochloride and Chemotherapy in Treating Patients With Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Sprint for Life (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0800; NCI-2012-00056 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-0800 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Undifferentiated Carcinoma; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Adenocarcinoma; Ovarian Undifferentiated Carcinoma; Primary Peritoneal Serous Adenocarcinoma; Stage II Fallopian Tube Cancer AJCC v6 and v7; Stage II Ovarian Cancer AJCC v6 and v7; Stage IIA Fallopian Tube Cancer AJCC v6 and v7; Stage IIA Ovarian Cancer AJCC V6 and v7; Stage IIB Fallopian Tube Cancer AJCC v6 and v7; Stage IIB Ovarian Cancer AJCC v6 and v7; Stage IIC Fallopian Tube Cancer AJCC v6 and v7; Stage IIC Ovarian Cancer AJCC v6 and v7; Stage III Fallopian Tube Cancer AJCC v7; Stage III Ovarian Cancer AJCC v6 and v7; Stage III Primary Peritoneal Cancer AJCC v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Drug Therapy; Propranolol; propranolol CR

ARMS (1):
- Treatment (propranolol hydrochloride) (Experimental): Patients receive propranolol hydrochloride PO BID beginning 48-72 hours before treatment. Patients undergoing surgery resume propranolol hydrochloride post-operatively once oral drugs are tolerated and continue until completion of 6 cycles of chemotherapy. Patients undergoing neoadjuvant chemotherapy continue propranolol hydrochloride PO BID during 3 chemotherapy cycles pre-surgery and 3 cycles post-surgery. Treatment repeats every 3 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Chemotherapy; Drug: Propranolol Hydrochloride; Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Chemotherapy — Undergo standard chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Drug: Propranolol Hydrochloride — Given PO
  Other Names: Inderal; Innopran XL
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection

SUMMARY:
This early phase I trial studies giving propranolol hydrochloride with standard chemotherapy in treating patients with ovarian, primary peritoneal, or fallopian tube cancer. Biological therapies, such as propranolol hydrochloride, blocks certain chemicals that affect the heart and this may stimulate the immune system and allow the chemotherapy to kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of pharmacologic beta-adrenergic blockade in women with stages II-IV epithelial ovarian cancer patients (n=25) either during initial tumor reductive surgery and through the first six cycles of standard intravenous chemotherapy or during neoadjuvant chemotherapy followed by surgery and further chemotherapy (chemo) up to a total of 6 cycles.

SECONDARY OBJECTIVES:

I. To characterize the biobehavioral states of these patients by using the Functional Assessment of Chronic Illness and Therapy- Ovary (FACT-O), Hospital Anxiety and Depression Survey (HADS) and the Center for Epidemiologic Studies Depression Scale (CESD) and serum levels of angiogenic cytokines at points pre- and post-treatment with beta-blockers.

II. To follow patients for progression-free survival (PFS) and overall survival (OS).

TRANSLATIONAL OBJECTIVES:

I. Determining vascular endothelial growth factor (VEGF), interleukin (IL)-6, IL-8, and other cytokines levels in patients with ovarian cancer who are receiving beta-blockers and comparing these levels pre-treatment and during treatment with response.

OUTLINE:

Patients receive propranolol hydrochloride orally (PO) twice daily (BID) beginning 48-72 hours before treatment. Patients undergoing surgery resume propranolol hydrochloride post-operatively once oral drugs are tolerated and continue until completion of 6 cycles of chemotherapy. Patients undergoing neoadjuvant chemotherapy continue propranolol hydrochloride PO BID during 3 chemotherapy cycles pre-surgery and 3 cycles post-surgery. Treatment repeats every 3 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Suspected preoperative diagnosis of invasive epithelial ovarian cancer, primary peritoneal carcinoma, fallopian tube cancer based on imaging and cancer antigen (Ca) 125; histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell carcinoma, mixed epithelial carcinoma, or adenocarcinoma not otherwise specified; patients with primarily carcinoma histology but mixed features can be included; the surgically confirmed histologic features must be compatible with primary Mullerian epithelial adenocarcinoma
* Stages II-IV of the above cancer
* Patients to be scheduled for a planned tumor debulking
* Intention for chemotherapy administration at MD Anderson Cancer Center
* Zubrod performance status 0-2
* Absolute neutrophil count (ANC) >= 1500/ml
* Platelets > 100,000/mL
* Creatinine clearance (CrCl) > 50 mL/min
* Bilirubin =< 1.5 x institutional upper limit normal
* Serum glutamic oxaloacetic transaminase (SGOT) =< 2.5 x institutional upper limit normal
* Alkaline phosphatase =< 2.5 x institutional upper limit normal
* Neuropathy (sensory and motor) =< grade 1 according to Common Toxicity Criteria for Adverse Events version 3 (CTCAE)
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin for the management of venous thrombosis including pulmonary embolus)
* Partial thromboplastin time (PTT) < 1.2 times institutional upper limit of normal
* Pulse >= 60 beat per minute (bpm)
* Systolic blood pressure (SBP) > 110 mmHg; diastolic blood pressure (DBP) >= 60 mmHg
* Normotensive individuals not already on beta blockers (may be on other anti hypertensives): SBP =< 140, DBP =< 90
* Surgery or neoadjuvant chemotherapy must be scheduled at least 72 hours in advance in order for the patient to take at least 48 hours of prescribed propranolol and have stable vital signs confirmed
* An approved informed consent and authorization permitting release of personal health information must be signed by patient or guardian
* Patients of childbearing age must have a negative pregnancy test
* Patients who receive neoadjuvant chemotherapy for their ovarian, primary peritoneal, or fallopian tube cancer

Exclusion Criteria:

* Patients with non-epithelial ovarian tumors that do not require adjuvant chemotherapy, borderline epithelial ovarian tumor, or recurrent invasive epithelial ovarian, low grade ovarian cancer, primary peritoneal, or fallopian tube cancer treated with surgery only (such as patients with stage IA or IB); patients with a prior diagnosis of a borderline tumor that was surgically resected and who subsequently develop an unrelated new invasive epithelial ovarian, primary peritoneal, or fallopian tube cancer are eligible, provided that they have not received chemotherapy for any tumor; no stromal cancers or germ cell cancers or low malignant potential; patients found post operatively to have ineligible histology will be removed from the study
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded; prior radiation therapy for localized cancer of the breast, head and neck, or skin is permitted provided that it was completed more than 3 years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients with a synchronous primary endometrial cancer, or a past history of primary endometrial cancer are excluded unless all of the following conditions are met: stage not greater than stage IA; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell, or other International Federation of Gynecology and Obstetrics (FIGO) grade 3 lesions
* Patients who have received targeted therapy (including but not limited to vaccines, antibodies, tyrosine kinase inhibitors) or hormonal therapy for management of their primary peritoneal, ovarian, or fallopian tube cancer
* With the exception of non-melanoma skin cancer and other specific malignancies as noted above, patients with other invasive malignancies who had (or have) any evidence of the other cancer present within the last five years or whose previous cancer treatment contraindicates this protocol therapy are excluded
* Metastases to the ovaries from other organs except fallopian tube or primary peritoneal carcinoma
* Use of systemic glucocorticoids such as prednisone or Decadron in the last month
* Inability to accurately answer questions (e.g. dementia, brain metastases) or speak English or Spanish
* Cirrhosis of the liver
* Patients with a Zubrod performance status 3 or 4
* Comorbid conditions: Addison's disease, autoimmune hepatitis, hepatitis B, hepatitis C, acquired immunodeficiency syndrome (AIDS) or human immunodeficiency virus (HIV), lupus erythematosus, mixed connective tissue disease, rheumatoid arthritis
* Any patients already on beta-blockers or contraindicated to receive beta-blockers
* Hypersensitivity to propranolol, or beta-blockers
* Uncompensated congestive heart failure
* Cardiogenic shock
* Severe sinus bradycardia; heart block, second or third degree or sick sinus syndrome (if no artificial pacemaker present)
* Severe hyperactive airway disease (chronic obstructive pulmonary disease, asthma)
* Any patients planning to receive Avastin or any other anti-angiogenic drugs
* Patients with brittle diabetes mellitus (DM); brittle diabetes mellitus is a type of diabetes when a person's blood glucose (sugar) level often swings quickly from high to low and from low to high; also called "unstable diabetes" or "labile diabetes"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03-09 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who successfully complete 6 cycles of chemotherapy with propranolol hydrochloride | Up to 6 months
  The success rate will be estimated with a 90% credible interval.

SECONDARY OUTCOMES:
Changes in quality of life as measured by the Functional Assessment of Chronic Illness and Therapy- Ovary (FACT-O) | Baseline to up to 6 months
  Descriptive statistics will be used to summarize measurements at each assessment time, and boxplots and histograms will be used to illustrate the distribution of this outcome at each assessment time. Changes from baseline will be similarly summarized. If these data are approximately normally distributed, or transformable to be approximately normally distributed, mixed repeated measures models and linear contrasts will be used to test for changes over time and associations between these quantities. Highly skewed measures analyzed using nonparametric methods.
Changes in mood state as measured by the Hospital Anxiety and Depression Survey (HADS) | Baseline to up to 6 months
  Descriptive statistics will be used to summarize measurements at each assessment time, and boxplots and histograms will be used to illustrate the distribution of this outcome at each assessment time. Changes from baseline will be similarly summarized. If these data are approximately normally distributed, or transformable to be approximately normally distributed, mixed repeated measures models and linear contrasts will be used to test for changes over time and associations between these quantities. Highly skewed measures analyzed using nonparametric methods.
Progression-free survival (PFS) | Up to 1 year
  PFS will be estimated with the product-limit estimator of Kaplan and Meier illustrated with a Kaplan-Meier plot. Proportional hazards models will be used to examine the association between cytokines and PFS.
Overall survival (OS) | Up to 1 year
  Will be estimated with the product-limit estimator of Kaplan and Meier. Proportional hazards models will be used to examine the association between cytokines and OS.
Incidence of adverse events | Up to 1 year after completion of study treatment
  Adverse events will be tabulated with particular attention to grade 3-4 neutropenia and grade 2+ neurotoxicity. The incidence of each type of adverse event will be estimated with a 95% confidence interval.
Changes in mood state as measured by Center for Epidemiologic Studies Depression Scale (CES-D | Baseline to up to 6 months
  scriptive statistics will be used to summarize measurements at each assessment time, and boxplots and histograms will be used to illustrate the distribution of this outcome at each assessment time. Changes from baseline will be similarly summarized. If these data are approximately normally distributed, or transformable to be approximately normally distributed, mixed repeated measures models and linear contrasts will be used to test for changes over time and associations between these quantities. Highly skewed measures analyzed using nonparametric methods.

OTHER OUTCOMES:
"Changes in immune response, measured by serum levels of IL-6 | Baseline to up to 6 months
  Descriptive statistics will be used to summarize measurements at each assessment time, and boxplots and histograms will be used to illustrate the distribution of this outcome at each assessment time. Changes from baseline will be similarly summarized. If these data are approximately normally distributed, or transformable to be approximately normally distributed, mixed repeated measures models and linear contrasts will be used to test for changes over time and associations between these quantities. Highly skewed measures analyzed using nonparametric methods.
Changes in immune response, measured by serum levels of IL-8 | Baseline to up to 6 months
  Descriptive statistics will be used to summarize measurements at each assessment time, and box-plots and histograms will be used to illustrate the distribution of this outcome at each assessment time. Changes from baseline will be similarly summarized. If these data are approximately normally distributed, or transformable to be approximately normally distributed, mixed repeated measures models and linear contrasts will be used to test for changes over time and associations between these quantities. Highly skewed measures analyzed using non-parametric methods.
Changes in immune response, measured by serum levels of VEGF | Baseline to up to 6 months
  Descriptive statistics will be used to summarize measurements at each assessment time, and boxplots and histograms will be used to illustrate the distribution of this outcome at each assessment time. Changes from baseline will be similarly summarized. If these data are approximately normally distributed, or transformable to be approximately normally distributed, mixed repeated measures models and linear contrasts will be used to test for changes over time and associations between these quantities. Highly skewed measures analyzed using non-parametric methods.

CONTACTS AND LOCATIONS:
Overall Officials: Lois M Ramondetta, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- United States (7):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - MD Anderson in Katy, Houston, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - MD Anderson in The Woodlands, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org